CLINICAL TRIAL: NCT01514097
Title: Adequacy of Pain Management for Upper Extremity Fracture After Discharge From a Pediatric Emergency Depart
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Children's Hospitals and Clinics of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1112-120
Record Dates: First submitted 2012-01-12; First posted 2012-01-20 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2014-04

CONDITIONS: Fracture
Keywords: emergency; pediatric; fracture; pain
MeSH Terms: conditions — Fractures, Bone; Emergencies; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Fractures reduced
- Fractures splinted

SUMMARY:
Pain is a common cause for children seeking care in the Emergency Department (ED). Children with orthopedic injuries often require pain control when seeking emergency care. Despite the high prevalence of ED visits requiring pain control, pain is often poorly assessed and treated in ED settings. Currently, no standard of care exists for the management of this fracture-related pain in children discharged from the ED. Furthermore, discrepancies in analgesia administration to patients of various racial groups seeking emergency care have been documented but are poorly understood. No research currently exists comparing pain severity between upper extremity fractures requiring simple splinting to those treated with sedated reduction and splinting. Furthermore, there is no research regarding the prevalence of significant post-discharge pain nor the differences among ethnic and age groups treated in the ED.

Research Questions:

What is the prevalence of significant post-discharge pain in children treated for upper extremity fractures?

Is there a difference in severity between those children requiring reduction versus simple splinting?

Is there a difference in pain severity noted among different ethnic or age groups?

Design This is a prospective, un-blinded, observational study that will include patients seeking treatment for an upper extremity fracture.

ELIGIBILITY:
Inclusion Criteria:

* Parents/guardians of patients presenting to the ED will be included if:
* The patient is younger than 18 years old
* The patient has an isolated upper extremity fracture (including clavicle, humerus, forearm, wrist) undergoing ED splinting with or without reduction
* The parent/guardian is English, Spanish, Somali, or Hmong-speaking
* The parent/guardian lives with the child
* He/she has a working telephone number

Exclusion Criteria:

* Potential subjects presenting to the ED will be excluded from study participation if:
* There is suspicion of child abuse or neglect
* The parent/guardian is not English, Spanish, Somali, or Hmong-speaking
* The patient is critically ill
* The fracture requires operative reduction/treatment
* The patient is medically complex
* The patient has a pre-existing bone disease or chronic pain syndrome

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric emergency department
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-02; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Pain Score | day 2 - 3
  Numeric pain scale from 0 - 10. 10 indicating the worst pain

SECONDARY OUTCOMES:
Second pain score assessment | 7-8 days after ED discharge
  Numeric pain scale from 0 - 10. 10 indicating the worst pain

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospitals and Clinics of Minnesota, Twin Cities, Minnesota, United States